CLINICAL TRIAL: NCT04256668
Title: Identification and Characterization of Human Sperm Variation and Its Role in Embryonic Development.
Brief Title: Human Sperm Epigenetics in Embryonic Development.
Acronym: EPI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Friedrich Miescher Institute for Biomedical Research (FMI) (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: Human Sperm Epigenetic
Record Dates: First submitted 2020-01-27; First posted 2020-02-05 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Male Infertility; Epigenetic Disorder
Keywords: assisted reproductive technology; DNA fragmentation; histone; protamine; blastocyst
MeSH Terms: conditions — Infertility, Male | interventions — Semen Analysis

STUDY DESIGN:
Intervention Model Description: 20 infertile men treated with assisted reproduction with normal embryo development in vitro, as demonstrated in a previous treatment with assisted reproductive technology (defined by normal fertilization rate >50% and normal blastocyst development rate >50%).
  20 infertile men treated with assisted reproduction with poor embryo development in vitro, as demonstrated in a previous treatment with assisted reproductive technology (defined by normal or slightly reduced fertilization rate <50% and low or absent blastocyst development (0 or only 1 blastocyst).
  20 previously infertile men, normal history, normal genital status, normal sperm count, DNA fragmentation rate <20% (as given by TUNEL) and achieving pregnancy naturally (without medical intervention).
Who Masked: Investigator, Outcomes Assessor
Masking Description: Sperm samples will be collected, processed and stained at the hospital site (RME). Slides generated for imaging will be assigned an anonymous code, removing all possible patient identifiable features. Then the slides will be sent to the research laboratory (FMI) for further analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- good embryo development in assisted reproduction (Active Comparator): 20 infertile men treated with assisted reproduction with normal embryo development in vitro, as demonstrated in a previous treatment with assisted reproductive technology (defined by normal fertilization rate >50% and normal blastocyst development rate >50%).
  Interventions: Diagnostic Test: Obtaining one or semen samples
- poor embryo development in assisted reproduction (Active Comparator): 20 infertile men treated with assisted reproduction with poor embryo development in vitro, as demonstrated in a previous treatment with assisted reproductive technology (defined by normal or slightly reduced fertilization rate <50% and low or absent blastocyst development (0 or only 1 blastocyst).
  Interventions: Diagnostic Test: Obtaining one or semen samples
- natural conception (Placebo Comparator): 20 previously infertile men, normal history, normal genital status, normal sperm count, DNA fragmentation rate <20% (as given by TUNEL) and achieving pregnancy naturally (without medical intervention).
  Interventions: Diagnostic Test: Obtaining one or semen samples

INTERVENTIONS:
Diagnostic Test: Obtaining one or semen samples — Through staining of semen samples with sets of dyes to measure features of chromatin density, nuclear morphology and mitochondrial status in large numbers of single spermatozoa and to compare differences in the staining results with known fertility outcome. Through comprehensive comparative epigenetic studies we anticipate to explain different efficiencies of sperm from men with seemingly normal semen quality in driving embryonic development.
  Other Names: Semen analysis

SUMMARY:
A total of 60 men (40 with a history of infertility and treatment with assisted reproduction and 20 infertile controls achieving conception naturally) will be asked to provide at least one semen sample each for conventional semen analysis including measurement of DNA-fragmentation and semen preparation with swim-up. The prepared semen sample will then analyzed by comprehensive microscopy analyses aiming at identifying distinct subpopulations of spermatozoa based on chromatin density and composition, mitochondrial and acrosome function and epigenetic markers. In addition, spermatozoa samples of selected individuals will be subjected to comprehensive analyses of the chromatin and RNA expression status using epigenomic approaches.

DETAILED DESCRIPTION:
Hitherto male infertility has been defined by conventional semen analysis only, which mainly consists of determining concentration, progressive mobility and morphology of spermatozoa. However, the diagnostic accuracy of conventional semen analysis is poor and has very limited relationship with the outcome of assisted reproductive medicine. Preliminary data suggest that differences in chromatin density and epigenetic status of sperm may be more relevant, in particular with respect to the growth and differentiation of early embryos.

Chromatin density, morphology, mitochondrial status and epigenetic state in sperm of infertile men with disturbances of early embryo development in vitro will be compared with those of infertile men with normal embryo development and with fertile controls.

Primary outcome:

Features of chromatin density will be determined through staining of large numbers of spermatozoa. Differences in the staining results will be compared with known fertility outcome.

Secondary outcome:

Development of significant staining parameters towards the selection against sperm with reduced embryonic competence and/or in favor of sperm supporting embryonic development after assisted reproduction, thereby using flow cytometry and sorting (FACS) .

ELIGIBILITY:
Inclusion Criteria:

* Men with a history of infertility. Sperm concentration must be >15 millions per ml.

Exclusion Criteria:

* No vulnerable persons will be invited to participate.

Ages: 28 Years to 39 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Differences in chromatin density. | 12 months
  Staining of the nucleus of spermatozoa with the fluorescent dye chromomycin

SECONDARY OUTCOMES:
Normal and abnormal embryo development after assisted reproduction. | 24 months
  Differences in distribution of epigenetic markers.

CONTACTS AND LOCATIONS:
Overall Officials: Christian De Geyter, MD, Principal Investigator — University Hospital
Locations (1):
- University Hospital, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gill ME, Fischer M, De Geyter C, Peters AHFM. Normozoospermic infertile men possess subpopulations of sperm varying in DNA accessibility, relating to differing reproductive outcomes. Hum Reprod. 2025 Jul 1;40(7):1266-1281. doi: 10.1093/humrep/deaf081. PMID 40375809